CLINICAL TRIAL: NCT01480180
Title: A Multi-national Trial Evaluating Safety and Efficacy, Including Pharmacokinetics, of NNC 0129-0000-1003 When Administered for Treatment and Prophylaxis of Bleeding in Patients With Haemophilia A
Brief Title: Evaluation of Safety and Efficacy, Including Pharmacokinetics, of NNC 0129-0000-1003 When Administered for Treatment and Prophylaxis of Bleeding in Subjects With Haemophilia A
Acronym: pathfinder™2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7088-3859; U1111-1119-7416 (Other: WHO); 2011-001142-15 (EudraCT Number); JapicCTI-121749 (Other: Japic)
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylaxis (Experimental)
  Interventions: Drug: turoctocog alfa pegol
- On-demand (Experimental)
  Interventions: Drug: turoctocog alfa pegol

INTERVENTIONS:
Drug: turoctocog alfa pegol — Administered i.v.
  Other Names: NNC 0129-0000-1003

SUMMARY:
This trial is conducted globally. The aim of the trial is to evaluate the safety and efficacy, including pharmacokinetics (the exposure of the trial drug in the body) of NNC 0129-0000-1003 (N8-GP) in subjects with Haemophilia A.

ELIGIBILITY:
Inclusion Criteria: - Male patients with severe congenital haemophilia A (FVIII activity below 1%, according to medical records) - Documented history of at least 150 EDs (exposure days) to other FVIII products - At least 12 years and body weight at least 35 kg (except for Croatia, France, Russia, Israel and the Netherlands where the lower age limit will be 18 years) Exclusion Criteria: - Previous participation in this trial defined as withdrawal after administration N8-GP - Any history of FVIII inhibitors - FVIII inhibitors above or equal to 0.6 BU/mL at screening - HIV (human immunodeficiency virus) positive, defined by medical records with CD4+ (T-lymphocyte subtype) count below or equal to 200/mcL or a viral load of more than 400000 copies/mL. If the data is not available in medical records within last 6 months, CD4+ will be measured at the screening visit - Congenital or acquired coagulation disorders other than haemophilia A - Previous significant thromboembolic events (e.g. myocardial infarction, cerebrovascular disease or deep venous thrombosis) as defined by available medical records - Platelet count below 50,000 platelets/mcL (laboratory value at the screening visit) - ALAT (alanine aminotransferase) above 3 times the upper limit of normal reference ranges at central laboratory - Creatinine level equal to or greater than 1.5 times above upper normal limit (according to central laboratory reference ranges) - Ongoing immune modulating or chemotherapeutic medication

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2012-01-30 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (88):
- United States (29):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, Torrance, California
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Boise, Idaho
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, East Lansing, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, New Brunswick, New Jersey
  - Novo Nordisk Investigational Site, Newark, New Jersey
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Charlottesville, Virginia
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
- Australia (3):
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, South Brisbane, Queensland
  - Novo Nordisk Investigational Site, Parkville, Victoria
- Novo Nordisk Investigational Site, Campinas, São Paulo, Brazil
- Novo Nordisk Investigational Site, Sofia, Bulgaria
- Croatia (2):
  - Novo Nordisk Investigational Site, Split
  - Novo Nordisk Investigational Site, Zagreb
- Denmark (2):
  - Novo Nordisk Investigational Site, Århus N
  - Novo Nordisk Investigational Site, København Ø
- France (4):
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Paris
- Germany (6):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Frankfurt/M.
  - Novo Nordisk Investigational Site, Hanover
  - Novo Nordisk Investigational Site, Homburg
  - Novo Nordisk Investigational Site, München
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
- Novo Nordisk Investigational Site, Tel Litwinsky, Israel
- Italy (4):
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Udine
  - Novo Nordisk Investigational Site, Vicenza
- Japan (9):
  - Novo Nordisk Investigational Site, Aichi
  - Novo Nordisk Investigational Site, Hiroshima
  - Novo Nordisk Investigational Site, Kitakyusyu, Fukuoka
  - Novo Nordisk Investigational Site, Nara
  - Novo Nordisk Investigational Site, Saitama
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shizuoka
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Yokohama-shi, Kanagawa
- Malaysia (2):
  - Novo Nordisk Investigational Site, Kuala Lumpur
  - Novo Nordisk Investigational Site, Selangor Darul Ehsan
- Netherlands (2):
  - Novo Nordisk Investigational Site, Groningen
  - Novo Nordisk Investigational Site, Rotterdam
- Novo Nordisk Investigational Site, Oslo, Norway
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- Novo Nordisk Investigational Site, Saint Petersburg, Russia
- Novo Nordisk Investigational Site, Daejeon, South Korea
- Spain (2):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
- Novo Nordisk Investigational Site, Malmo, Sweden
- Switzerland (3):
  - Novo Nordisk Investigational Site, Geneva
  - Novo Nordisk Investigational Site, Lausanne
  - Novo Nordisk Investigational Site, Zurich
- Taiwan (2):
  - Novo Nordisk Investigational Site, Changhua
  - Novo Nordisk Investigational Site, Taipei
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, Samsun
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Basingstoke
  - Novo Nordisk Investigational Site, Cardiff
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Sheffield

REFERENCES:
- [Result] Giangrande P, Chowdary P, Enhrenforth S, Hanabusa H, Leebeek FW, Lentz SR, Nemes L, Poulsen LH, Santagostino E, You CW, Clausen WHO, Oldenburg J and on behalf of for the pathfinder™2 Investigators. Clinical evaluation of novel recombinant glycopegylated FVIII (turoctocog alfa pegol, N8-GP): efficacy and safety in previously treated patients with severe hemophilia A - results of pathfinder™2 international trial. Journal of Thrombosis and Haemostasis (Abstracts) 2015; 13 (Supplement S2): 1-997 [OR212]
- [Result] Giangrande P, Andreeva T, Chowdary P, Ehrenforth S, Hanabusa H, Leebeek FW, Lentz SR, Nemes L, Poulsen LH, Santagostino E, You CW, Clausen WH, Jonsson PG, Oldenburg J; Pathfinder2 Investigators. Clinical evaluation of glycoPEGylated recombinant FVIII: Efficacy and safety in severe haemophilia A. Thromb Haemost. 2017 Jan 26;117(2):252-261. doi: 10.1160/TH16-06-0444. Epub 2016 Dec 1. PMID 27904904
- [Result] Giangrande P, Abdul Karim F, Nemes L, You CW, Landorph A, Geybels MS, Curry N. Long-term safety and efficacy of N8-GP in previously treated adults and adolescents with hemophilia A: Final results from pathfinder2. J Thromb Haemost. 2020 Sep;18 Suppl 1(Suppl 1):5-14. doi: 10.1111/jth.14959. PMID 32544297
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 77 sites in 22 countries as follows: Australia:3; Brazil:1; Croatia:1; Denmark:2; France:3; Germany:5; Hungary:2; Israel:1; Italy:2; Japan:8; Malaysia:2; Netherlands:2; Norway:1; Russian Federation:1; Korea, Republic of:1; Spain:2; Sweden:1; Switzerland:3; Taiwan:2; Turkey:3; United Kingdom:6; United States:25.
Pre-assignment Details: The trial had a main phase and an extension phase 1 and phase 2.
Groups:
- Prophylaxis: Participants received one single bolus dose of 50 U/kg of body weight (BW) of turoctocog alfa pegol (N8-GP), administered intravenously (IV) every 4th day (96 hours) or twice weekly (investigator's discretion). The dose was based on phase 1 data from the NN7088-3776 trial in order to ensure a trough level of >1% FVIII:C activity in the majority of participants in the prophylaxis arm. This arm is applicable only for the main phase.
- On-demand: Participants received treatment with N8-GP in case of a bleeding episode. All bleeds were to be treated with doses between 20-75 U/kg BW according to the severity and location of the bleeding episode. The dosage (N8-GP units) was calculated by multiplying the participant's weight in kilograms by the desired factor level multiplied by 0.5. This arm is applicable only for the main phase.
- N8-GP 50 U/kg Prophylaxis Q4D: Participants who were on prophylaxis treatment with N8-GP in the main phase and had 0-2 bleeding episodes during the last 6 months before entering the extension phase, were included in this arm. Participants received one single bolus dose of 50 U/kg BW of N8-GP administered IV every 4th day (96 hours) or twice weekly (at investigator's discretion). The dose was adjusted to ensure a trough level of >1% FVIII:C activity in this arm. The dose was based on phase 1 data from the NN7088-3776 trial in order to ensure a trough level of >1% FVIII:C activity in the majority of participants in the prophylaxis arm. This arm was applicable for the extension phase part-1 and part 2.
- N8-GP 75 U/kg Prophylaxis Q7D: Participants who were on prophylaxis treatment with N8-GP in the main phase and had 3+ bleeding episodes during the last 6 months before entering the extension phase, were randomised to receive one single bolus dose of 75 U/kg BW of N8-GP. Participants received one single bolus dose of 75 U/kg BW of N8-GP administered IV every 7th day (Q7D). Based on the bleeding pattern, the investigator could change the dosing frequency from Q7D to Q4D, but not vice versa. The dose was based on phase 1 data from the NN7088-3776 trial in order to ensure a trough level of >1% FVIII:C activity in the majority of participants in the prophylaxis arm.
- N8-GP 20-75 U/kg On-demand: Participants received treatment with N8-GP in case of a bleeding episode. All bleeds were to be treated with doses between 20-75 U/kg BW according to the severity and location of the bleeding episode. The dosage (N8-GP units) was calculated by multiplying the participant's weight in kilograms by the desired factor level multiplied by 0.5.
- N8-GP Prophylaxis: Participants in this arm include subjects both from the 50 U/kg Q4D and the 75 U/kg Q7D prophylaxis arms.
Period: Main Phase
Arm/Group | Prophylaxis | On-demand | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand | N8-GP Prophylaxis
Started | 174 | 12 | 0 (Not applicable for this phase) | 0 (Not applicable for this phase) | 0 (Not applicable for this phase) | 0 (Not applicable for this phase)
Max. Participants After Switching | 175 | 11 | 0 | 0 | 0 | 0
Completed | 155 | 11 | 0 (Not applicable for this phase) | 0 (Not applicable for this phase) | 0 (Not applicable for this phase) | 0 (Not applicable for this phase)
Not Completed | 19 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal criteria | 12 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Unclassified | 3 | 0 | 0 | 0 | 0 | 0
Period: Extension Phase, Part 1
Arm/Group | Prophylaxis | On-demand | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand | N8-GP Prophylaxis
Started | 0 | 0 | 105 | 38 | 7 | 0
Completed | 0 | 0 | 95 | 28 | 7 | 0
Not Completed | 0 | 0 | 10 | 10 | 0 | 0
Not completed — Withdrawal criteria | 0 | 0 | 5 | 0 | 0 | 0
Not completed — Unclassified | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 4 | 1 | 0 | 0
Not completed — Change of treatment | 0 | 0 | 0 | 9 | 0 | 0
Period: Extension Phase, Part 2
Arm/Group | Prophylaxis | On-demand | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand | N8-GP Prophylaxis
Started | 0 | 0 | 94 | 40 | 5 | 0
Completed | 0 | 0 | 77 | 33 | 3 | 0
Not Completed | 0 | 0 | 17 | 7 | 2 | 0
Not completed — Withdrawal criteria | 0 | 0 | 10 | 6 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Unclassified | 0 | 0 | 3 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prophylaxis: Participants received one single bolus dose of 50 U/kg of body weight (BW) of turoctocog alfa pegol (N8-GP), administered intravenously (IV) every 4th day (96 hours) or twice weekly (investigator's discretion). The dose was based on phase 1 data from the NN7088-3776 trial in order to ensure a trough level of >1% FVIII:C activity in the majority of participants in the prophylaxis arm.
- On-demand: Participants received treatment with N8-GP in case of a bleeding episode. All bleeds were to be treated with doses between 20-75 U/kg BW according to the severity and location of the bleeding episode. The dosage (N8-GP units) was calculated by multiplying the participant's weight in kilograms by the desired factor level multiplied by 0.5.
- Total: Total of all reporting groups
Arm/Group | Prophylaxis | On-demand | Total
Number analyzed (Participants) | 174 | 12 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (12.4) | 39.8 (13.9) | 31.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 174 | 12 | 186
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity of participants
  Participants
    Hispanic or Latino | 13 | 0 | 13
    Not Hispanic or Latino | 161 | 12 | 173
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race of the participants
  Participants
    Asian | 31 | 4 | 35
    Black or African American | 8 | 3 | 11
    White | 133 | 5 | 138
    Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Incidence Rate of FVIII-inhibitors ≥0.6 BU: After Approximately 19 Months
Description: All participants with neutralizing antibodies were included in the numerator and any participant with a minimum 50 exposure days plus any participant with inhibitory inhibitors was included in the denominator. A positive inhibitor test was defined as ≥0.6 bethesda unit (BU). Estimates are based on exact calculations for a binomial distribution. For the calculation of the 'inhibitor rate' the nominator included all participants with neutralising antibodies while the denominator included all participants with a minimum of 50 exposures plus any participant with less than 50 exposures but with neutralising inhibitors.
Time Frame: After approximately 19 months
Population: Results are based on the safety analysis set (SAS). SAS comprised all participants exposed to N8-GP in this trial. Number analysed = Number of participants with available data for respective arm.
Measure: Number; unit: Inhibitor rate
Groups:
- N8-GP 50 U/kg Prophylaxis Q4D: Participants received one single bolus dose of 50 U/kg of body weight (BW) of N8-GP administered intravenously (IV) every 4th day (96 hours) or twice weekly (investigator's discretion). The dose was based on phase 1 data from the NN7088-3776 trial in order to ensure a trough level of >1% FVIII:C activity in the majority of participants in the prophylaxis arm.
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Inhibitor rate | 0.006 | 0

2. Primary Outcome: Annualised Bleeding Rate in the Prophylaxis Arm: After Approximately 19 Months
Description: Annualised bleeding rate (ABR) is the number of bleeding episodes per year. This was assessed only for the prophylaxis treatment with N8-GP.
Time Frame: After approximately 19 months
Population: Results were based on the full analysis set (FAS) which included all participants exposed to N8-GP in this trial. Number analysed = Number of participants with available data for respective arm.
Measure: Median (Inter-Quartile Range); unit: Bleeds per participant per year
Groups:
- N8-GP Prophylaxis: Participants from both the N8-GP 50 U/kg Q4D and N8-GP 75 U/kg Q7D groups were included in this arm.
Arm/Group | N8-GP Prophylaxis
Number analyzed (Participants) | 177
Bleeds per participant per year | 1.33 [0 to 4.61]
Statistical Analysis 1: Comparison: N8-GP Prophylaxis; The analysis is based on a Poisson regression model allowing for over-dispersion. For participants withdrawing prematurely, the log planned treatment duration is used as offset; for completers, the log actual treatment duration is used; Test type: Other; p < 0.001, Poisson regression — P-values are from the 1-sided test of the null hypothesis that the ABR is at least 8.5 evaluated at the 2.5% level; Poisson estimate = 3.70, 95% CI 2-sided [2.94 to 4.66]

3. Primary Outcome: The Incidence Rate of FVIII-inhibitors ≥0.6 BU: After Approximately 25 Months
Description: as for outcome 1
Time Frame: After approximately 25 months
Population: Results are based on the SAS. SAS comprised all participants exposed to N8-GP in this trial. Number analysed = Number of participants with available data for respective arm.
Measure: Number; unit: Inhibitor rate
Groups:
- N8-GP 50 U/kg Prophylaxis Q4D: Participants who were on prophylaxis treatment with N8-GP in the main phase and had 0-2 bleeding episodes during the last 6 months before entering the extension phase, were included in this arm. Participants received one single bolus dose of 50 U/kg BW of N8-GP administered IV every 4th day (96 hours) or twice weekly (at investigator's discretion). The dose was adjusted to ensure a trough level of >1% FVIII:C activity in this arm. The dose was based on phase 1 data from the NN7088-3776 trial in order to ensure a trough level of >1% FVIII:C activity in the majority of participants in the prophylaxis arm.
- N8-GP 20-75 U/kg On-demand: Participants in this arm received treatment with N8-GP in case of a bleeding episode. All bleeds were to be treated with doses between 20-75 U/kg BW according to the severity and location of the bleeding episode. The dosage (N8-GP units) was calculated by multiplying the participant's weight in kilograms by the desired factor level multiplied by 0.5.
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
Inhibitor rate | 0.006 | 0 | 0

4. Primary Outcome: Annualised Bleeding Rate in the Prophylaxis Arm: After Approximately 25 Months
Description: ABR is the number of bleeding episodes per year. This was assessed only for the prophylaxis treatment with N8-GP.
Time Frame: After approximately 25 months
Population: Results are based on the FAS which included all participants exposed to N8-GP in this trial. Number analysed = Number of participants with available data for respective arm.
Measure: Median (Inter-Quartile Range); unit: Bleeds per participant per year
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D
Number analyzed (Participants) | 177 | 61
Bleeds per participant per year | 1.36 [0.00 to 4.00] | 0 [0.00 to 2.36]
Statistical Analysis 1: Comparison: N8-GP 50 U/kg Prophylaxis Q4D; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Poisson regression — P-values are from the 1-sided test of the null hypothesis that the ABR is at least 8.5 evaluated at the 2.5% level; Poisson estimate = 3.27, 95% CI 2-sided [2.59 to 4.11]

5. Primary Outcome: Incidence Rate of FVIII-inhibitors ≥0.6 BU: At Approximately 80 Months
Description: as for outcome 1
Time Frame: At approximately 80 months
Population: as for outcome 3
Measure: Number; unit: Inhibitor rate
Arm/Group | N8-GP Prophylaxis | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Inhibitor rate | 0.006 | 0

6. Primary Outcome: Annualised Bleeding Rate in the Prophylaxis Arm: After Approximately 80 Months
Description: Annualised bleeding rate (ABR) is the number of bleeding episodes per year reported during the prophylactic treatment with N8-GP.
Time Frame: After approximately 80 months
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial. Number analysed = Number of participants with available data for respective arm.
Measure: Median (Inter-Quartile Range); unit: Bleeds per participant per year
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D
Number analyzed (Participants) | 177 | 61
Bleeds per participant per year | 0.99 [0.00 to 2.68] | 1.95 [0.43 to 6.52]
Statistical Analysis 1: Comparison: N8-GP 50 U/kg Prophylaxis Q4D; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Poisson regression — P-values are from the 1-sided test of the null hypothesis that the ABR is at least 8.5 evaluated at the 2.5% level; Poisson estimate = 2.35, 95% CI 2-sided [1.87 to 2.95]
Statistical Analysis 2: Comparison: N8-GP 75 U/kg Prophylaxis Q7D; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Poisson regression — P-values are from the 1-sided test of the null hypothesis that the ABR is at least 8.5 evaluated at the 2.5% level; Poisson estimate = 4.39, 95% CI 2-sided [3.09 to 6.24]

7. Secondary Outcome: Haemostatic Effect of N8-GP When Used for Treatment of Bleeds, Assessed on a Four-point Scale for Haemostatic Response (Excellent, Good, Moderate and None): After Approximately 19 Months
Description: Haemostatic effect of N8-GP for treatment of bleeding episodes was assessed by 4-point response scale: none, moderate, good or excellent. Evaluation during trial was done by participant and/or parent(s)/caregiver within approximately 8 hours after a single injection as follows: Excellent: Abrupt pain relief and/or clear improvement in objective signs of bleeding within approximately 8 hrs after a single injection; Good: Definite pain relief and/or improvement in signs of bleeding within approximately 8 hrs after a single injection, but possibly requiring more than one injection for complete resolution; Moderate: Probable or slight beneficial effect within approximately 8 hours after the first injection, but usually requiring more than one injection; None: No improvement, or worsening of symptoms.
Time Frame: After approximately 19 months
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial. Number analysed = Number of bleeds analysed.
Measure: Count of Units; unit: Bleeding episodes
Units Other Than Participants: Bleeding episodes
Groups:
- N8-GP 20-75 U/kg On-demand: Participants who were on prophylaxis treatment with N8-GP in the main phase and had 3+ bleeding episodes during the last 6 months before entering the extension phase, were randomised to receive one single bolus dose of 75 U/kg BW of N8-GP. Participants received one single bolus dose of 75 U/kg BW of N8-GP administered IV every 7th day (Q7D). Based on the bleeding pattern, the investigator could change the dosing frequency from Q7D to Q4D, but not vice versa. The dose was based on phase 1 data from the NN7088-3776 trial in order to ensure a trough level of >1% FVIII:C activity in the majority of participants in the prophylaxis arm.
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 175 | 12
Number analyzed (Bleeding episodes) | 436 | 532
Bleeding episodes
  Excellent | 192 | 320
  Good | 174 | 170
  Moderate | 62 | 41
  None | 4 | 1
  Missing | 4 | 0

8. Secondary Outcome: Haemostatic Effect of N8-GP When Used for Treatment of Bleeds, Assessed on a Four-point Scale for Haemostatic Response (Excellent, Good, Moderate and None): After Approximately 25 Months
Description: as for outcome 7
Time Frame: After approximately 25 months
Population: as for outcome 7
Measure: Count of Units; unit: Bleeding episodes
Units Other Than Participants: Bleeding episodes
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
Number analyzed (Bleeding episodes) | 716 | 25 | 695
Bleeding episodes
  Excellent | 330 | 9 | 406
  Good | 270 | 11 | 233
  Moderate | 98 | 3 | 55
  None | 4 | 0 | 1
  Missing | 14 | 2 | 0

9. Secondary Outcome: Haemostatic Effect of N8-GP When Used for Treatment of Bleeds, Assessed on a Four-point Scale for Haemostatic Response (Excellent, Good, Moderate and None): After Approximately 80 Months
Description: as for outcome 7
Time Frame: After approximately 80 months
Population: as for outcome 7
Measure: Count of Units; unit: Bleeding episodes
Units Other Than Participants: Bleeding episodes
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
Number analyzed (Bleeding episodes) | 1312 | 176 | 1270
Bleeding episodes
  Excellent | 600 | 75 | 859
  Good | 532 | 65 | 339
  Moderate | 153 | 29 | 71
  None | 6 | 2 | 1
  Missing | 21 | 5 | 0

10. Secondary Outcome: Consumption of N8-GP Per Bleeding Episode (Number of Infusions): After Approximately 19 Months
Description: The mean number of infusions of N8-GP used for treatment of a bleed from start to stop of a bleed was reported.
Time Frame: After approximately 19 months
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial. Number analysed = Number of infusions in respective arm.
Measure: Mean (Standard Deviation); unit: Number of infusions
Units Other Than Participants: Infusions
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Number analyzed (Infusions) | 436 | 532
Number of infusions | 1.4 (1.0) | 1.2 (0.9)

11. Secondary Outcome: Consumption of N8-GP Per Bleeding Episode (Number of Infusions): After Approximately 25 Months
Description: The mean number of infusions of N8-GP used for treatment of a bleed from start to stop of a bleed was reported.
Time Frame: After approximately 25 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Number of infusions
Units Other Than Participants: Infusions
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
Number analyzed (Infusions) | 716 | 25 | 695
Number of infusions | 1.4 (1.3) | 1.3 (0.6) | 1.2 (0.8)

12. Secondary Outcome: Consumption of N8-GP Per Bleeding Episode (Number of Infusions): After Approximately 80 Months
Description: The mean number of infusions of N8-GP used for treatment of a bleed from start to stop of a bleed was reported.
Time Frame: After approximately 80 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Number of infusions
Units Other Than Participants: Infusions
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
Number analyzed (Infusions) | 1312 | 176 | 1270
Number of infusions | 1.4 (1.3) | 1.3 (0.6) | 1.2 (0.8)

13. Secondary Outcome: Consumption of N8-GP Per Bleeding Episode (U/kg): After Approximately 19 Months
Description: The mean consumption of N8-GP (U/kg) used for treatment of a bleed from start to stop of a bleed was reported.
Time Frame: After approximately 19 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/kg per bleed
Units Other Than Participants: Bleeding episodes
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Number analyzed (Bleeding episodes) | 436 | 532
U/kg per bleed | 64.6 (48.8) | 41.0 (35.1)

14. Secondary Outcome: Consumption of N8-GP Per Bleeding Episode (U/kg): After Approximately 25 Months
Description: The mean consumption of N8-GP (U/kg) used for treatment of a bleed from start to stop of a bleed was reported.
Time Frame: After approximately 25 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/kg per bleed
Units Other Than Participants: Bleeding episodes
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
Number analyzed (Bleeding episodes) | 716 | 25 | 695
U/kg per bleed | 67.8 (72.9) | 78.2 (37.8) | 39.3 (32.4)

15. Secondary Outcome: Consumption of N8-GP Per Bleeding Episode (U/kg): After Approximately 80 Months
Description: The mean consumption of N8-GP (U/kg) used for treatment of a bleed from start to stop of a bleed was reported.
Time Frame: After approximately 80 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/kg per bleed
Units Other Than Participants: Bleeding episodes
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
Number analyzed (Bleeding episodes) | 1310 | 175 | 1270
U/kg per bleed | 68.1 (60.0) | 88.7 (72.4) | 37.5 (38.0)

16. Secondary Outcome: Consumption of N8-GP (Number of Infusions) During Prophylaxis and On-demand Treatment: After Approximately 19 Months
Description: Number of infusions are presented as average dose used during propphylaxis and on-demand treatment.
Time Frame: After approximately 19 months
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial. Number analysed = Number of infusions used during prophylaxis and on-demand treatment.
Measure: Mean (Standard Deviation); unit: U/kg
Units Other Than Participants: Infusions
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Number analyzed (Infusions) | 436 | 532
U/kg | 52.2 (1.4) | 46.3 (10.4)

17. Secondary Outcome: Consumption of N8-GP (Number of Infusions) During Prophylaxis and On-demand Treatment: After Approximately 25 Months
Description: Number of infusions are presented as average dose used during prophylaxis and on-demand treatment.
Time Frame: After approximately 25 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: U/kg
Units Other Than Participants: Infusions
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 175 | 38 | 12
Number analyzed (Infusions) | 22569 | 775 | 35
U/kg | 52.2 (1.9) | 77.2 (3.2) | 44.8 (11.4)

18. Secondary Outcome: Consumption of N8-GP (Number of Infusions) During Prophylaxis and On-demand Treatment: After Approximately 80 Months
Description: Number of infusions are presented as average dose used during prophylaxis and on-demand treatment.
Time Frame: After approximately 80 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: U/kg
Units Other Than Participants: Infusions
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
Number analyzed (Infusions) | 55896 | 6996 | 58
U/kg | 52.2 (1.5) | 77.1 (3.2) | 37.5 (13.0)

19. Secondary Outcome: Consumption of N8-GP (U/kg Per Month) During Prophylaxis and On-demand Treatment: After Approximately 19 Months
Description: The mean consumption of N8-GP used for treatment of a bleed from start to stop of a bleed (per month per participant) was reported.
Time Frame: After approximately 19 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/kg per month
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
U/kg per month | 403.8 (53.8) | 129.2 (71.8)

20. Secondary Outcome: Consumption of N8-GP (U/kg Per Month) During Prophylaxis and On-demand Treatment: After Approximately 25 Months
Description: as for outcome 19
Time Frame: After approximately 25 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/kg per month
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
U/kg per month | 403.8 (53.8) | 349.2 (37.9) | 128.2 (70.1)

21. Secondary Outcome: Consumption of N8-GP (U/kg Per Month) During Prophylaxis and On-demand Treatment: After Approximately 80 Months
Description: as for outcome 19
Time Frame: After approximately 80 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/kg per month
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
U/kg per month | 402.4 (52.4) | 353.5 (32.9) | 130.2 (69.2)

22. Secondary Outcome: Consumption of N8-GP (U/kg Per Year) During Prophylaxis and On-demand Treatment: After Approximately 19 Months
Description: The mean consumption of N8-GP used for treatment of a bleed from start to stop of a bleed (per year per participant) was reported.
Time Frame: After approximately 19 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/kg per year
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
U/kg per year | 4845 (645) | 1550 (861)

23. Secondary Outcome: Consumption of N8-GP (U/kg Per Year) During Prophylaxis and On-demand Treatment: After Approximately 25 Months
Description: as for outcome 22
Time Frame: After approximately 25 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/kg per year
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
U/kg per year | 4846 (645.3) | 4190 (454.5) | 1538 (840.6)

24. Secondary Outcome: Consumption of N8-GP (U/kg Per Year) During Prophylaxis and On-demand Treatment: After Approximately 80 Months
Description: as for outcome 22
Time Frame: After approximately 80 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/kg per year
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
U/kg per year | 4829 (628.8) | 4242 (394.5) | 1562 (830.3)

25. Secondary Outcome: Haemostatic Effect as Measured by Recovery and Trough Levels FVIII:C (in All Patients Receiving Prophylaxis Treatment): After Approximately 19 Months
Description: Recovery and trough levels of FVIII:C was reported for all participants at Visit 3 (Week 4) and end of main phase (approx. 19 months). The data was reported for all participants who received prophylaxis treatment. Chromogenic assay was performed with N8-GP product specific standard (PSS) as a calibrator.
Time Frame: After approximately 19 months
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/mL
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D
Number analyzed (Participants) | 177
U/mL
  Visit 2 Post-dose: number analyzed (Participants) | 168
  Visit 2 Post-dose | 1.276 (18.584)
  Visit 3 Pre-dose: number analyzed (Participants) | 148
  Visit 3 Pre-dose | 0.030 (159.920)
  Visit 12 Post-dose: number analyzed (Participants) | 46
  Visit 12 Post-dose | 1.359 (18.156)
  Visit 13 Pre-dose: number analyzed (Participants) | 143
  Visit 13 Pre-dose | 0.034 (188.891)

26. Secondary Outcome: Haemostatic Effect as Measured by Recovery and Trough Levels FVIII:C (in All Patients Receiving Prophylaxis Treatment): After Approximately 25 Months
Description: Recovery and trough levels of FVIII:C was reported for all participants at the end of extension phase 1 study (approx. 25 months). The data was reported for all participants who received prophylaxis treatment. Chromogenic assay was performed with N8-GP product specific standard (PSS) as a calibrator.
Time Frame: After approximately 25 months
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/mL
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D
Number analyzed (Participants) | 177 | 61
U/mL
  Visit 16 Post-dose: number analyzed (Participants) | 15 | 30
  Visit 16 Post-dose | 1.329 (13.357) | 1.868 (31.919)
  Visit 17 Pre-dose: number analyzed (Participants) | 16 | 28
  Visit 17 Pre-dose | 0.028 (205.652) | 0.015 (272.494)

27. Secondary Outcome: Haemostatic Effect as Measured by Recovery and Trough Levels FVIII:C (in All Patients Receiving Prophylaxis Treatment): After Approximately 80 Months
Description: Since patients were allowed to change prophylaxis regimen at any time during the extension phase part 2, and since the visit intervals were different for the 2 prophylaxis treatment regimens (Q4D and Q7D), FVIII activity data are reported only as incremental recovery at this timepoint.
Time Frame: After approximately 80 months
Population: Data were not collected for this endpoint.
Groups:
- N8-GP 75 U/kg Prophylaxis Q7D: Participants in this arm received treatment with N8-GP in case of a bleeding episode. All bleeds were to be treated with doses between 20-75 U/kg BW according to the severity and location of the bleeding episode. The dosage (N8-GP units) was calculated by multiplying the participant's weight in kilograms by the desired factor level multiplied by 0.5.
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Patient Reported Outcomes - Change in HAEMO-QOL Total Scores (Patients 13-16 Years Old) After Approx 19 and 25 Months
Description: Reported results are change from baseline (Month 0) measured at end of main phase (approx Month 19) and change from Month 19 at end of Extension 1 (approx Month 25) of the study. The HAEMO-QOL assessment included questions on physical health, feeling, view of yourself, family, friends, perceived support, other persons, sports and school, dealing with haemophilia, treatment, future, and relationships. Scores range for each question was 0-100, with a lower score indicating better quality of life related to haemophilia.
Time Frame: After approx 19 and 25 months
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial. Number analysed = Number of participants with available data. No participants from the 13-16 years age group received on-demand treatment. Thus on-demand treatment group is not applicable for this endpoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- N8-GP 50 U/kg Prophylaxis Q4D: Participants from the N8-GP 50 U/kg Q4D group were included in this arm.
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D
Number analyzed (Participants) | 16
Scores on a scale
  Approx month 19 (Change from baseline): number analyzed (Participants) | 10
  Approx month 19 (Change from baseline) | -0.1 (12.4)
  Approx month 25 (Change from month 19): number analyzed (Participants) | 7
  Approx month 25 (Change from month 19) | 0.8 (4.5)

29. Secondary Outcome: Patient Reported Outcomes - Change in HAEMO-QOL Total Scores (Patients 13-16 Years Old): After Approx 80 Months
Description: Reported results are change from visit 1 (Month 0) upto end of Extension phase 2 (Month 80) of the study. Time intervals are assigned based on time after first dose. It was possible that a participant could answer more than one questionnaire in a single time interval. The HAEMO-QOL assessment included questions on physical health, feeling, view of yourself, family, friends, perceived support, other persons, sports and school, dealing with haemophilia, treatment, future, and relationships. Scores range for each question was 0-100, with a lower score indicating better quality of life related to haemophilia. Overall number of units analysed = Maximum no of questionnaires answered by participants for this endpoint. Overall number of participants analysed = maximum number of participants contributed to the analysis for each time point.
Time Frame: 2-<3 yrs, 3-<4 yrs, 4-<5 yrs, 5-<6 yrs and 6-<7 yrs
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial. No participants from the 13-16 years age group received on-demand treatment. Thus on-demand treatment group is not applicable for this endpoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Number of questionnaires
Groups:
- N8-GP Prophylaxis: Participants from both the 50 U/kg Q4D and the 75 U/kg Q7D prophylaxis arms were included in this arm.
Arm/Group | N8-GP Prophylaxis
Number analyzed (Participants) | 11
Number analyzed (Number of questionnaires) | 11
Scores on a scale
  2 to <3 years (Change from baseline): number analyzed (Number of questionnaires) | 6
  2 to <3 years (Change from baseline) | 2.7 (15.9)
  3 to <4 years (Change from baseline): number analyzed (Number of questionnaires) | 8
  3 to <4 years (Change from baseline) | -0.9 (11.6)
  4 to <5 years (Change from baseline): number analyzed (Number of questionnaires) | 10
  4 to <5 years (Change from baseline) | 2.6 (15.8)
  5 to <6 years (Change from baseline) | 2.1 (11.7)
  6 to <7 years (Change from baseline): number analyzed (Number of questionnaires) | 1
  6 to <7 years (Change from baseline) | -0.3 (0)

30. Secondary Outcome: Patient Reported Outcomes - Change in HAEMO-QOL Total Scores (Parents of Patients 13-16 Years Old): After Approx 19 and 25 Months
Description: Reported results are change from baseline (Month 0) measured at end of main phase (Month 19) and change from Month 19 to end of Extension 1 (Month 25) of the study. The questionnaire was completed by parents of the patients in the 13-16 years old age bracket. The HAEMO-QOL assessment included questions on physical health, feeling, view of yourself, family, friends, perceived support, other persons, sports and school, dealing with haemophilia, treatment, future, and relationships. Scores range for each question was 0-100, with a lower score indicating better quality of life related to haemophilia.
Time Frame: After approx 19 and 25 months
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D
Number analyzed (Participants) | 16
Scores on a scale
  After approximately 19 months: number analyzed (Participants) | 9
  After approximately 19 months | -4.0 (13.1)
  After approximately 25 months: number analyzed (Participants) | 6
  After approximately 25 months | 1.8 (8.3)

31. Secondary Outcome: Patient Reported Outcomes - Change in HAEMO-QOL Total Scores (Parents of Patients 13-16 Years Old): After Approx 80 Months
Description: Reported results are change from visit 1 (Month 0) upto end of Extension phase 2 (Month 80) of the study. The questionnaire was completed by parents of the patients in the 13-16 years old age bracket. Time intervals are assigned based on time after first dose. It was possible that a participant could answer more than one questionnaire in a single time interval. The HAEMO-QOL assessment included questions on physical health, feeling, view of yourself, family, friends, perceived support, other persons, sports and school, dealing with haemophilia, treatment, future, and relationships. Scores range for each question was 0-100, with a lower score indicating better quality of life related to haemophilia. Overall number of units analysed = Maximum no of questionnaires answered by participants for this endpoint. Overall number of participants analysed = maximum number of participants contributed to the analysis for each time point.
Time Frame: 2-<3 yrs, 3-<4 yrs, 4-<5 yrs, 5-<6 yrs and 6-<7 yrs
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Number of questionnaires
Arm/Group | N8-GP Prophylaxis
Number analyzed (Participants) | 9
Number analyzed (Number of questionnaires) | 8
Scores on a scale
  2 to <3 years (Change from baseline): number analyzed (Number of questionnaires) | 6
  2 to <3 years (Change from baseline) | 1.5 (2.1)
  3 to <4 years (Change from baseline): number analyzed (Number of questionnaires) | 7
  3 to <4 years (Change from baseline) | -8.1 (7.0)
  4 to <5 years (Change from baseline) | -7.9 (13.8)
  5 to <6 years (Change from baseline) | 1.6 (11.4)
  6 to <7 years (Change from baseline): number analyzed (Number of questionnaires) | 1
  6 to <7 years (Change from baseline) | 10.7 (0)

32. Secondary Outcome: Patient Reported Outcomes - Change in HAEM-A-QOL (>=17 Years) Total Scores: After Approx 19 and 25 Months
Description: Reported results are change from baseline (Month 0) measured at end of main phase (Month 19) and change from Month 19 to end of Extension 1 (Month 25) of the study. The HAEM-A-QOL (for adults (>=17 years)) assessment included questions on questions on physical health, feeling, view of yourself, sports and leisure, work and school, dealing with haemophilia, treatment, future, family planning, and partnership and sexuality. Scores range for each question was 0-100, with a lower score indicating better quality of life related to haemophilia.
Time Frame: After approx 19 and 25 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 157 | 12
Scores on a scale
  Week 76 (Change from baseline): number analyzed (Participants) | 154 | 11
  Week 76 (Change from baseline) | -2.3 (8.9) | -3.1 (10.3)
  Week 140 (Change from week 76): number analyzed (Participants) | 113 | 6
  Week 140 (Change from week 76) | 0.7 (8.0) | -0.6 (4.9)

33. Secondary Outcome: Patient Reported Outcomes - Change in HAEM-A-QOL (>=17 Years) Total Scores: After Approximately 80 Months
Description: Reported results are change from visit 1 (Month 0) upto end of Extension phase 2 (Month 80) of the study. Time intervals are assigned based on time after first dose. It was possible that a participant could answer more than one questionnaire in a single time interval. Overall number of units analysed = Maximum no of questionnaires answered by participants for this endpoint. Overall number of participants analysed = maximum number of participants contributed to the analysis for each time point. The HAEM-A-QOL (for adults (>=17 years)) assessment included questions on physical health, feeling, view of yourself, sports and leisure, work and school, dealing with haemophilia, treatment, future, family planning, and partnership and sexuality. Scores range for each question was 0-100, with a lower score indicating better quality of life related to haemophilia. Scores range for each question was 0-100, with a lower score indicating better quality of life related to haemophilia.
Time Frame: 2-<3 yrs, 3-<4 yrs, 4-<5 yrs, 5-<6 yrs and 6-<7 yrs
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Number of questionnaires
Arm/Group | N8-GP Prophylaxis | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 122 | 5
Number analyzed (Number of questionnaires) | 157 | 5
Scores on a scale
  1 to <2 years (Change from baseline): number analyzed (Participants) | 122 | 0
  1 to <2 years (Change from baseline): number analyzed (Number of questionnaires) | 9 | 0
  1 to <2 years (Change from baseline) | -6.6 (6.7) |
  2 to <3 years (Change from baseline): number analyzed (Number of questionnaires) | 118 | 2
  2 to <3 years (Change from baseline) | -2.6 (10.3) | -10.7 (8.7)
  3 to <4 years (Change from baseline): number analyzed (Number of questionnaires) | 124 | 5
  3 to <4 years (Change from baseline) | -2.3 (8.9) | -5.8 (12.2)
  4 to <5 years (Change from baseline): number analyzed (Number of questionnaires) | 130 | 4
  4 to <5 years (Change from baseline) | -3.1 (10.4) | -2.5 (19.5)
  5 to <6 years (Change from baseline): number analyzed (Number of questionnaires) | 157 | 3
  5 to <6 years (Change from baseline) | -3.1 (11.2) | -1.7 (2.8)
  6 to <7 years (Change from baseline): number analyzed (Number of questionnaires) | 22 | 4
  6 to <7 years (Change from baseline) | -3.5 (9.0) | -7.8 (8.6)

34. Secondary Outcome: Patient Reported Outcomes - Change in HEMO-SAT (Patients) Scores: After Approx 19 and 25 Months
Description: Reported results are change from baseline (Month 0) measured at end of main phase (Month 19) and change from Month 19 to end of Extension 1 (Month 25) of the study. The HEMO-SAT (Hematology-satisfaction) assessment included questions on treatment aspects including Ease and convenience, efficacy, burden, specialist/nurses, centre/hospital, general satisfaction (reported by patients). Adults completing the questionnaire could achieve a score from 0 to 100, with lower scores reflecting greater treatment satisfaction. The scale range for each of the 6 domains was 0-100 with lower scores reflecting greater treatment satisfaction. A decrease in the score would mean improvement.
Time Frame: After approx 19 and 25 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 157 | 12
Scores on a scale
  Ease & convenience (Change - Approx 19 months): number analyzed (Participants) | 152 | 10
  Ease & convenience (Change - Approx 19 months) | -0.4 (13.8) | -4.5 (11.5)
  Ease & convenience (Change - Approx 25 months): number analyzed (Participants) | 113 | 6
  Ease & convenience (Change - Approx 25 months) | 0.3 (11.7) | -6.3 (6.9)
  Efficacy (Change - Approx 19 months): number analyzed (Participants) | 151 | 10
  Efficacy (Change - Approx 19 months) | -6.3 (15.6) | -11.3 (11.1)
  Efficacy (Change - Approx 25 months): number analyzed (Participants) | 114 | 6
  Efficacy (Change - Approx 25 months) | -0.2 (11.0) | 0.0 (5.9)
  Burden (Change - Approx 19 months): number analyzed (Participants) | 152 | 10
  Burden (Change - Approx 19 months) | -2.2 (15.8) | -5.0 (18.8)
  Burden (Change - Approx 25 months): number analyzed (Participants) | 114 | 6
  Burden (Change - Approx 25 months) | -0.9 (11.3) | 0.0 (6.3)
  Speciaist/nurses (Change - approx 19 months): number analyzed (Participants) | 152 | 11
  Speciaist/nurses (Change - approx 19 months) | -2.9 (11.7) | -4.5 (8.3)
  Speciaist/nurses (Change - approx 25 months): number analyzed (Participants) | 114 | 6
  Speciaist/nurses (Change - approx 25 months) | 1.8 (9.1) | 0.0 (8.1)
  Centre/hospital (Change - approx 19 months): number analyzed (Participants) | 151 | 11
  Centre/hospital (Change - approx 19 months) | -2.2 (11.9) | -3.6 (7.8)
  Centre/hospital (Change - approx 25 months): number analyzed (Participants) | 114 | 6
  Centre/hospital (Change - approx 25 months) | 1.0 (8.1) | 4.2 (10.7)
  Gen. satisfaction (Change - approx 19 months): number analyzed (Participants) | 151 | 11
  Gen. satisfaction (Change - approx 19 months) | -2.9 (15.4) | -3.4 (11.3)
  Gen. satisfaction (Change - approx 25 months): number analyzed (Participants) | 113 | 6
  Gen. satisfaction (Change - approx 25 months) | -1.1 (9.4) | 2.1 (5.1)

35. Secondary Outcome: Patient Reported Outcomes - Change in HEMO-SAT (Patients) Scores: After Approximately 80 Months
Description: Reported results are change from visit 1 (Month 0) upto end of Extension phase 2 (Month 80) of the study. Time intervals are assigned based on time after first dose. It was possible that a participant could answer more than one questionnaire in a single time interval. Overall number of units analysed = Maximum no of questionnaires answered by participants for this endpoint. Overall number of participants analysed = maximum number of participants contributed to the analysis for each time point. The HEMO-SAT assessment included questions on treatment aspects including Ease and convenience, efficacy, burden, specialist/nurses, centre/hospital, general satisfaction (reported by patients). Adults completing the questionnaire could achieve a score from 0 to 100, with lower scores reflecting greater treatment satisfaction. The scale range for each of the 6 domains was 0-100 with lower scores reflecting greater treatment satisfaction. A decrease in the score would mean improvement.
Time Frame: 1-<2 yrs, 2-<3 yrs, 3-<4 yrs, 4-<5 yrs, 5-<6 yrs and 6-<7 yrs
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Number of questionnaires
Arm/Group | N8-GP Prophylaxis | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 122 | 5
Number analyzed (Number of questionnaires) | 151 | 5
Scores on a scale
  Ease & convenience 1 to <2 years: number analyzed (Number of questionnaires) | 9 | 0
  Ease & convenience 1 to <2 years | -2.2 (12.7) |
  Ease & convenience 2 to <3 years: number analyzed (Number of questionnaires) | 117 | 2
  Ease & convenience 2 to <3 years | -2.4 (14.4) | -23.8 (12.4)
  Ease & convenience 3 to <4 years: number analyzed (Number of questionnaires) | 124 | 5
  Ease & convenience 3 to <4 years | -3.7 (13.6) | -10.5 (18.3)
  Ease & convenience 4 to <5 years: number analyzed (Number of questionnaires) | 120 | 4
  Ease & convenience 4 to <5 years | -3.7 (13.6) | -4.4 (34.4)
  Ease & convenience 5 to <6 years: number analyzed (Number of questionnaires) | 151 | 3
  Ease & convenience 5 to <6 years | -3.3 (13.7) | -16.7 (11.8)
  Ease & convenience 6 to <7 years: number analyzed (Number of questionnaires) | 21 | 4
  Ease & convenience 6 to <7 years | -7.2 (12.4) | -5.6 (8.3)
  Efficacy 1 to <2 years: number analyzed (Number of questionnaires) | 9 | 0
  Efficacy 1 to <2 years | -1.9 (9.3) |
  Efficacy 2 to <3 years: number analyzed (Number of questionnaires) | 117 | 2
  Efficacy 2 to <3 years | -7.1 (14.9) | -16.7 (5.9)
  Efficacy 3 to <4 years: number analyzed (Number of questionnaires) | 124 | 5
  Efficacy 3 to <4 years | -7.2 (13.6) | -17.5 (14.3)
  Efficacy 4 to <5 years: number analyzed (Number of questionnaires) | 119 | 4
  Efficacy 4 to <5 years | -9.5 (16.4) | 2.1 (35.8)
  Efficacy 5 to <6 years: number analyzed (Number of questionnaires) | 150 | 3
  Efficacy 5 to <6 years | -7.4 (14.4) | -16.7 (20.8)
  Efficacy 6 to <7 years: number analyzed (Number of questionnaires) | 21 | 4
  Efficacy 6 to <7 years | -13.2 (21.8) | -3.1 (13.8)
  Burden 1 to <2 years: number analyzed (Number of questionnaires) | 9 | 0
  Burden 1 to <2 years | 0.7 (13.4) |
  Burden 2 to <3 years: number analyzed (Number of questionnaires) | 117 | 2
  Burden 2 to <3 years | -3.6 (16.9) | -21.9 (4.4)
  Burden 3 to <4 years: number analyzed (Number of questionnaires) | 124 | 5
  Burden 3 to <4 years | -5.0 (15.1) | -17.5 (14.9)
  Burden 4 to <5 years: number analyzed (Number of questionnaires) | 119 | 4
  Burden 4 to <5 years | -4.9 (16.9) | -3.1 (28.2)
  Burden 5 to <6 years: number analyzed (Number of questionnaires) | 150 | 3
  Burden 5 to <6 years | -4.9 (13.5) | -18.8 (10.8)
  Burden 6 to <7 years: number analyzed (Number of questionnaires) | 21 | 4
  Burden 6 to <7 years | -10.1 (19.1) | -4.7 (9.4)
  Specialist/nurses 1 to <2 years: number analyzed (Number of questionnaires) | 9 | 0
  Specialist/nurses 1 to <2 years | -2.0 (12.8) |
  Specialist/nurses 2 to <3 years: number analyzed (Number of questionnaires) | 116 | 2
  Specialist/nurses 2 to <3 years | -2.8 (11.4) | 0.0 (0.0)
  Specialist/nurses 3 to <4 years: number analyzed (Number of questionnaires) | 124 | 5
  Specialist/nurses 3 to <4 years | -2.3 (10.9) | 0.7 (8.9)
  Specialist/nurses 4 to <5 years: number analyzed (Number of questionnaires) | 120 | 4
  Specialist/nurses 4 to <5 years | -1.4 (11.4) | 21.4 (47.7)
  Specialist/nurses 5 to <6 years: number analyzed (Number of questionnaires) | 150 | 3
  Specialist/nurses 5 to <6 years | -0.8 (9.7) | -11.9 (8.2)
  Specialist/nurses 6 to <7 years: number analyzed (Number of questionnaires) | 21 | 4
  Specialist/nurses 6 to <7 years | -0.2 (15.4) | -6.3 (7.4)
  Centre/hospital 1 to <2 years: number analyzed (Number of questionnaires) | 9 | 0
  Centre/hospital 1 to <2 years | -5.0 (12.0) |
  Centre/hospital 2 to <3 years: number analyzed (Number of questionnaires) | 116 | 2
  Centre/hospital 2 to <3 years | -2.9 (11.9) | 0.0 (0.0)
  Centre/hospital 3 to <4 years: number analyzed (Number of questionnaires) | 123 | 5
  Centre/hospital 3 to <4 years | -1.3 (10.5) | 3.0 (4.5)
  Centre/hospital 4 to <5 years: number analyzed (Number of questionnaires) | 118 | 4
  Centre/hospital 4 to <5 years | -1.1 (12.5) | 26.3 (43.1)
  Centre/hospital 5 to <6 years: number analyzed (Number of questionnaires) | 148 | 3
  Centre/hospital 5 to <6 years | -1.0 (9.7) | 1.7 (29.3)
  Centre/hospital 6 to <7 years: number analyzed (Number of questionnaires) | 21 | 4
  Centre/hospital 6 to <7 years | 1.2 (17.7) | -8.8 (6.3)
  Gen. satisfaction 1 to <2 years: number analyzed (Number of questionnaires) | 9 | 0
  Gen. satisfaction 1 to <2 years | -1.4 (11.6) |
  Gen. satisfaction 2 to <3 years: number analyzed (Number of questionnaires) | 117 | 2
  Gen. satisfaction 2 to <3 years | -4.1 (15.2) | -6.3 (8.8)
  Gen. satisfaction 3 to <4 years: number analyzed (Number of questionnaires) | 123 | 5
  Gen. satisfaction 3 to <4 years | -2.8 (10.7) | -17.5 (14.3)
  Gen. satisfaction 4 to <5 years: number analyzed (Number of questionnaires) | 119 | 4
  Gen. satisfaction 4 to <5 years | -5.0 (14.4) | 0.0 (35.4)
  Gen. satisfaction 5 to <6 years: number analyzed (Number of questionnaires) | 150 | 3
  Gen. satisfaction 5 to <6 years | -2.2 (12.2) | -20.8 (7.2)
  Gen. satisfaction 6 to <7 years: number analyzed (Number of questionnaires) | 21 | 4
  Gen. satisfaction 6 to <7 years | -5.4 (19.6) | -18.8 (16.1)

36. Secondary Outcome: Patient Reported Outcomes - Change in HEMO-SAT Scores (Parents): After Approx 19 and 25 Months
Description: The summary of change was based on individual changes observed at visit 13 (approximately 19 months) from visit 2a pre-dose (Month 0). The HEMO-SAT assessment included questions on treatment aspects including Ease and convenience, efficacy, burden, specialist/nurses, centre/hospital, general satisfaction (reported by parents). Adults completing the questionnaire could achieve a score from 0 to 100, with lower scores reflecting greater treatment satisfaction. The scale range for each of the 6 domains was 0-100 with lower scores reflecting greater treatment satisfaction. A decrease in the score would mean improvement.
Time Frame: After approx 19 and 25 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D
Number analyzed (Participants) | 16
Scores on a scale
  Ease & convenience - baseline (Week 0): number analyzed (Participants) | 10
  Ease & convenience - baseline (Week 0) | 27.8 (15.5)
  Ease & convenience (Change - Approx 19 months): number analyzed (Participants) | 9
  Ease & convenience (Change - Approx 19 months) | 0.4 (3.3)
  Ease & convenience (Change - Approx 25 months): number analyzed (Participants) | 7
  Ease & convenience (Change - Approx 25 months) | -6.3 (8.1)
  Efficacy - baseline (Week 0): number analyzed (Participants) | 10
  Efficacy - baseline (Week 0) | 17.9 (12.3)
  Efficacy (Change - Approx 19 months): number analyzed (Participants) | 9
  Efficacy (Change - Approx 19 months) | -5.2 (2.1)
  Efficacy (Change - Approx 25 months): number analyzed (Participants) | 7
  Efficacy (Change - Approx 25 months) | 2.1 (5.7)
  Burden- baseline (Week 0): number analyzed (Participants) | 10
  Burden- baseline (Week 0) | 23.8 (14.4)
  Burden (Change - Approx 19 months): number analyzed (Participants) | 9
  Burden (Change - Approx 19 months) | -10.9 (12.9)
  Burden (Change - Approx 25 months): number analyzed (Participants) | 7
  Burden (Change - Approx 25 months) | -4.2 (11.6)
  Specialist/nurses (Week 0): number analyzed (Participants) | 10
  Specialist/nurses (Week 0) | 7.1 (10.9)
  Speciaist/nurses (Change - approx 19 months): number analyzed (Participants) | 9
  Speciaist/nurses (Change - approx 19 months) | 0.0 (0.0)
  Speciaist/nurses (Change - approx 25 months): number analyzed (Participants) | 7
  Speciaist/nurses (Change - approx 25 months) | 0.6 (1.5)
  Centre/Hospital (Week 0): number analyzed (Participants) | 10
  Centre/Hospital (Week 0) | 10.5 (11.7)
  Centre/hospital (Change - approx 19 months): number analyzed (Participants) | 9
  Centre/hospital (Change - approx 19 months) | -3.7 (4.8)
  Centre/hospital (Change - approx 25 months): number analyzed (Participants) | 7
  Centre/hospital (Change - approx 25 months) | -0.8 (2.0)
  Gen. satisfaction (Week 0): number analyzed (Participants) | 10
  Gen. satisfaction (Week 0) | 8.8 (11.9)
  Gen. satisfaction (Change - approx 19 months): number analyzed (Participants) | 9
  Gen. satisfaction (Change - approx 19 months) | 0.0 (0.0)
  Gen. satisfaction (Change - approx 25 months): number analyzed (Participants) | 7
  Gen. satisfaction (Change - approx 25 months) | 0.0 (0.0)

37. Secondary Outcome: Patient Reported Outcomes - Change in HEMO-SAT (Parents) Scores: After Approximately 80 Months
Description: Reported results are from Visit 1 (Month 0), and change from visit 1 upto end of Extension phase 2 (Month 80) of the study. Time intervals are assigned based on time after first dose. It was possible that a participant could answer more than one questionnaire in a single time interval. Overall number of units analysed = Max. no of questionnaires answered by participants for this endpoint. Overall number of participants analysed = max. number of participants contributed to the analysis for each time point. The HEMO-SAT assessment included questions on treatment aspects including Ease and convenience, efficacy, burden, specialist/nurses, centre/hospital, general satisfaction. Adults completing the questionnaire could achieve a score from 0 to 100, with lower scores reflecting greater treatment satisfaction. The scale range for each of the 6 domains was 0-100 with lower scores reflecting greater treatment satisfaction. A decrease in the score would mean improvement.
Time Frame: 2-<3 yrs, 3-<4 yrs, 4-<5 yrs, 5-<6 yrs and 6-<7 yrs
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Number of questionnaires
Arm/Group | N8-GP Prophylaxis
Number analyzed (Participants) | 11
Number analyzed (Number of questionnaires) | 8
Scores on a scale
  Ease & convenience 2 to <3 years: number analyzed (Number of questionnaires) | 6
  Ease & convenience 2 to <3 years | -0.6 (6.8)
  Ease & convenience 3 to <4 years: number analyzed (Number of questionnaires) | 1
  Ease & convenience 3 to <4 years | 9.1 (0)
  Ease & convenience 4 to <5 years | -5.3 (14.1)
  Ease & convenience 5 to <6 years: number analyzed (Number of questionnaires) | 5
  Ease & convenience 5 to <6 years | -3.6 (13.5)
  Ease & convenience 6 to <7 years: number analyzed (Number of questionnaires) | 1
  Ease & convenience 6 to <7 years | 0.0 (0.0)
  Efficacy 2 to <3 years: number analyzed (Number of questionnaires) | 6
  Efficacy 2 to <3 years | -6.3 (2.4)
  Efficacy 3 to <4 years: number analyzed (Number of questionnaires) | 1
  Efficacy 3 to <4 years | -8.3 (0.0)
  Efficacy 4 to <5 years | -6.3 (4.4)
  Efficacy 5 to <6 years: number analyzed (Number of questionnaires) | 5
  Efficacy 5 to <6 years | 3.3 (17.0)
  Efficacy 6 to <7 years: number analyzed (Number of questionnaires) | 1
  Efficacy 6 to <7 years | -4.2 (0)
  Burden 2 to <3 years: number analyzed (Number of questionnaires) | 6
  Burden 2 to <3 years | -20.3 (15.6)
  Burden 3 to <4 years: number analyzed (Number of questionnaires) | 1
  Burden 3 to <4 years | -25.0 (0)
  Burden 4 to <5 years | -6.3 (26.2)
  Burden 5 to <6 years: number analyzed (Number of questionnaires) | 5
  Burden 5 to <6 years | 2.5 (15.1)
  Burden 6 to <7 years: number analyzed (Number of questionnaires) | 1
  Burden 6 to <7 years | -31.3 (0)
  Specialist/nurses 2 to <3 years: number analyzed (Number of questionnaires) | 6
  Specialist/nurses 2 to <3 years | -3.6 (7.1)
  Specialist/nurses 3 to <4 years: number analyzed (Number of questionnaires) | 1
  Specialist/nurses 3 to <4 years | 0.0 (0.0)
  Specialist/nurses 4 to <5 years | -6.5 (11.8)
  Specialist/nurses 5 to <6 years: number analyzed (Number of questionnaires) | 5
  Specialist/nurses 5 to <6 years | 3.6 (17.5)
  Specialist/nurses 6 to <7 years: number analyzed (Number of questionnaires) | 1
  Specialist/nurses 6 to <7 years | 0.0 (0.0)
  Centre/hospital 2 to <3 years: number analyzed (Number of questionnaires) | 6
  Centre/hospital 2 to <3 years | -3.7 (4.8)
  Centre/hospital 3 to <4 years: number analyzed (Number of questionnaires) | 1
  Centre/hospital 3 to <4 years | -5.0 (0.0)
  Centre/hospital 4 to <5 years | -8.3 (8.8)
  Centre/hospital 5 to <6 years: number analyzed (Number of questionnaires) | 5
  Centre/hospital 5 to <6 years | -3.0 (14.4)
  Centre/hospital 6 to <7 years: number analyzed (Number of questionnaires) | 1
  Centre/hospital 6 to <7 years | 0.0 (0.0)
  Gen. satisfaction 2 to <3 years: number analyzed (Number of questionnaires) | 6
  Gen. satisfaction 2 to <3 years | -9.4 (12.0)
  Gen. satisfaction 3 to <4 years: number analyzed (Number of questionnaires) | 1
  Gen. satisfaction 3 to <4 years | -12.5 (0)
  Gen. satisfaction 4 to <5 years | -6.3 (10.5)
  Gen. satisfaction 5 to <6 years: number analyzed (Number of questionnaires) | 5
  Gen. satisfaction 5 to <6 years | 5.0 (14.3)
  Gen. satisfaction 6 to <7 years: number analyzed (Number of questionnaires) | 1
  Gen. satisfaction 6 to <7 years | 0.0 (0.0)

38. Secondary Outcome: Patient Reported Outcomes - Change in EQ-5D-VAS Scores: After Approx 19 and 25 Months
Description: Reported results are change from baseline (Month 0) measured at end of main phase (Month 19) and change from Month 19 to end of Extension 1 (Month 25) of the study. The European quality of life visual analogue scale (EQ5D-VAS) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement. EQ-5D-VAS: range 0 to 100. A higher score indicates better self reported health status. A positive change indicates an improvement.
Time Frame: After approx 19 and 25 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 173 | 12
Scores on a scale
  Week 0 (Baseline): number analyzed (Participants) | 168 | 11
  Week 0 (Baseline) | 76.5 (17.9) | 74.5 (13.1)
  Week 76 (Change from baseline): number analyzed (Participants) | 159 | 11
  Week 76 (Change from baseline) | 2.0 (11.1) | 4.1 (7.2)
  Week 140 (Change from week 76): number analyzed (Participants) | 125 | 6
  Week 140 (Change from week 76) | -0.8 (11.8) | 2.7 (11.0)

39. Secondary Outcome: Patient Reported Outcomes - Change in EQ-5D-VAS Scores: After Approximately 80 Months
Description: Reported results are change from visit 1 (Month 0) upto end of Extension phase 2 (Month 80) of the study. Time intervals are assigned based on time after first dose. It was possible that a participant could answer more than one questionnaire in a single time interval. Overall number of units analysed = Maximum no of questionnaires answered by participants for this endpoint. Overall number of participants analysed = maximum number of participants contributed to the analysis for each time point. The EQ5D-VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement. EQ-5D-VAS: range 0 to 100. A higher score indicates better self reported health status. A positive change indicates an improvement.
Time Frame: 1-<2 yrs, 2-<3 yrs, 3-<4 yrs, 4-<5 yrs, 5-<6 yrs and 6-<7 yrs
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Number of questionnaires
Arm/Group | N8-GP Prophylaxis | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 133 | 5
Number analyzed (Number of questionnaires) | 167 | 5
Scores on a scale
  1 to <2 years (Change from baseline): number analyzed (Participants) | 133 | 0
  1 to <2 years (Change from baseline): number analyzed (Number of questionnaires) | 9 | 0
  1 to <2 years (Change from baseline) | 4.9 (8.2) |
  2 to <3 years (Change from baseline): number analyzed (Number of questionnaires) | 128 | 2
  2 to <3 years (Change from baseline) | 2.6 (13.3) | 9.5 (6.4)
  3 to <4 years (Change from baseline): number analyzed (Number of questionnaires) | 130 | 5
  3 to <4 years (Change from baseline) | 3.0 (13.5) | 7.3 (7.0)
  4 to <5 years (Change from baseline): number analyzed (Number of questionnaires) | 137 | 4
  4 to <5 years (Change from baseline) | 1.0 (15.8) | 11.0 (9.6)
  5 to <6 years (Change from baseline): number analyzed (Number of questionnaires) | 167 | 3
  5 to <6 years (Change from baseline) | 2.2 (13.2) | 15.0 (21.2)
  6 to <7 years (Change from baseline): number analyzed (Number of questionnaires) | 23 | 4
  6 to <7 years (Change from baseline) | 7.5 (13.6) | 16.3 (12.1)

40. Secondary Outcome: Patient Reported Outcomes - Change in European Quality of Life Utility Index: After Approx 19 and 25 Months
Description: Reported results are change from baseline (Month 0) measured at end of main phase (Month 19) and change from Month 19 to end of Extension 1 (Month 25) of the study. The European quality of life utility index comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels where 1 indicates better health state (no problems) and 3 indicates worst health state (confined to bed). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; a positive change indicates an improvement.
Time Frame: After approx 19 and 25 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 173 | 12
Scores on a scale
  Month 19 (Change from baseline): number analyzed (Participants) | 160 | 11
  Month 19 (Change from baseline) | 0.011 (0.184) | -0.028 (0.047)
  Month 25 (Change from Month 19): number analyzed (Participants) | 120 | 6
  Month 25 (Change from Month 19) | -0.025 (0.174) | -0.028 (0.093)

41. Secondary Outcome: Patient Reported Outcomes - Change in European Quality of Life Utility Index Scores: After Approximately 80 Months
Description: Reported results are change from visit 1 (Month 0) upto end of Extension phase 2 (Month 80) of the study. Time intervals are assigned based on time after first dose. It is possible that a patient answers more than one questionnaire in a single time interval. Overall units analysed = Max no. of questionnaires answered by participants for this endpoint. Overall no. of participants analysed = max no. of participants analysed at each time point. This utility index has 5 dimensions: mobility, self-care, usual activities, pain/discomfort & anxiety/depression. Each dimension has 3 levels where 1 indicates better health state (no problems) and 3 indicates worst health state (confined to bed). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; a positive change indicates an improvement.
Time Frame: 1-<2 yrs, 2-<3 yrs, 3-<4 yrs, 4-<5 yrs, 5-<6 yrs and 6-<7 yrs
Population: Results were based on the FAS which included all participants exposed to N8-GP in this trial.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Number of questionnaires
Arm/Group | N8-GP Prophylaxis | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 133 | 5
Number analyzed (Number of questionnaires) | 164 | 5
Scores on a scale
  1 to <2 years (Change from baseline): number analyzed (Number of questionnaires) | 9 | 0
  1 to <2 years (Change from baseline) | 0.052 (0.252) |
  2 to <3 years (Change from baseline): number analyzed (Number of questionnaires) | 128 | 2
  2 to <3 years (Change from baseline) | -0.008 (0.159) | 0.000 (0.000)
  3 to <4 years (Change from baseline): number analyzed (Number of questionnaires) | 130 | 5
  3 to <4 years (Change from baseline) | 0.021 (0.193) | 0.000 (0.000)
  4 to <5 years (Change from baseline): number analyzed (Number of questionnaires) | 139 | 4
  4 to <5 years (Change from baseline) | 0.000 (0.165) | -0.001 (0.057)
  5 to <6 years (Change from baseline): number analyzed (Number of questionnaires) | 164 | 3
  5 to <6 years (Change from baseline) | 0.011 (0.178) | 0.000 (0.000)
  6 to <7 years (Change from baseline): number analyzed (Number of questionnaires) | 23 | 4
  6 to <7 years (Change from baseline) | -0.062 (0.163) | 0.000 (0.000)

42. Secondary Outcome: Number of Hospital Admissions During the Trial
Description: The number of hospital admissions that took place in the study were reported.
Time Frame: After approx 19, 25 and 80 months
Population: as for outcome 6
Measure: Count of Units; unit: Number of hospital admissions
Units Other Than Participants: Number of hospital admissions
Arm/Group | N8-GP Prophylaxis | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 175 | 12
Number analyzed (Number of hospital admissions) | 110 | 12
Number of hospital admissions
  After approximately 19 months: number analyzed (Number of hospital admissions) | 52 | 8
  After approximately 19 months: 0 | 49 | 8
  After approximately 19 months: 1 | 3 | 0
  After approximately 19 months: 2 | 0 | 0
  After approximately 25 months: number analyzed (Number of hospital admissions) | 89 | 10
  After approximately 25 months: 0 | 84 | 8
  After approximately 25 months: 1 | 4 | 2
  After approximately 25 months: 2 | 1 | 0
  Month 25 to Month 80: number analyzed (Participants) | 134 | 5
  Month 25 to Month 80: number analyzed (Number of hospital admissions) | 21 | 2
  Month 25 to Month 80: 0 | 20 | 2
  Month 25 to Month 80: 1 | 1 | 0
  Month 25 to Month 80: 2 | 0 | 0

43. Secondary Outcome: Number of Days at the Hospital During the Trial
Description: The mean number of days that participants spent at the hospital during the study were reported.
Time Frame: After approx 19, 25 and 80 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | N8-GP Prophylaxis | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Days
  After approximately 19 months: number analyzed (Participants) | 52 | 8
  After approximately 19 months | 0.1 (0.4) | 0.0 (0.0)
  After approximately 25 months: number analyzed (Participants) | 89 | 10
  After approximately 25 months | 0.5 (3.8) | 0.7 (1.6)
  Month 25 to 80: number analyzed (Participants) | 21 | 2
  Month 25 to 80 | 0.5 (2.4) | 0.0 (0.0)

44. Secondary Outcome: Number of Admissions to the Emergency Room (ER) During the Trial
Description: The number of admissions to the ER that took place in the study were reported for each group.
Time Frame: After approx 19, 25 and 80 months
Population: as for outcome 6
Measure: Count of Units; unit: ER admissions
Units Other Than Participants: ER admissions
Arm/Group | N8-GP Prophylaxis | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 175 | 12
Number analyzed (ER admissions) | 110 | 12
ER admissions
  After approximately 19 months: number analyzed (ER admissions) | 52 | 8
  After approximately 19 months: 0 | 49 | 8
  After approximately 19 months: 1 | 1 | 0
  After approximately 19 months: 2 | 2 | 0
  After approximately 19 months: 4 | 0 | 0
  After approximately 25 months: number analyzed (ER admissions) | 89 | 10
  After approximately 25 months: 0 | 84 | 8
  After approximately 25 months: 1 | 2 | 1
  After approximately 25 months: 2 | 2 | 1
  After approximately 25 months: 4 | 1 | 0
  Month 25 to 80: number analyzed (Participants) | 134 | 5
  Month 25 to 80: number analyzed (ER admissions) | 21 | 2
  Month 25 to 80: 0 | 17 | 2
  Month 25 to 80: 1 | 4 | 0
  Month 25 to 80: 2 | 0 | 0
  Month 25 to 80: 4 | 0 | 0

45. Secondary Outcome: Number of Days Missing School or Work
Description: The mean number of days that participants missed to go to school or work were reported.
Time Frame: Approx 19, 25 and 80 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | N8-GP Prophylaxis | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Days
  After approximately 19 months: number analyzed (Participants) | 139 | 11
  After approximately 19 months | 0.5 (1.6) | 6.7 (16.9)
  After approximately 25 months: number analyzed (Participants) | 140 | 11
  After approximately 25 months | 0.8 (2.0) | 6.8 (16.9)
  Month 25 to 80: number analyzed (Participants) | 66 | 2
  Month 25 to 80 | 2.6 (14.4) | 0.3 (0.4)

46. Secondary Outcome: Number of Days Using Mobility Aid
Description: The mean number of days that participants used any aids for mobility during the study were reported.
Time Frame: Approx 19, 25 and 80 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | N8-GP Prophylaxis | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Days
  After approximately 24 months: number analyzed (Participants) | 162 | 12
  After approximately 24 months | 4.4 (26.2) | 11.1 (34.7)
  After approximately 36 months: number analyzed (Participants) | 165 | 12
  After approximately 36 months | 7.0 (42.7) | 5.8 (15.9)
  Month 25 to 80: number analyzed (Participants) | 77 | 2
  Month 25 to 80 | 1.0 (4.6) | 0.5 (0.7)

47. Secondary Outcome: Number of Participants Using Pain Medication
Description: The number of participants using pain medication during the main plus extension phase 1 of the study (approximately 25 months) and during extension phase 2(approximately 80 months) were reported.
Time Frame: After approx 25 and 80 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- N8-GP Prophylaxis: Participants in this arm included participants from both the Q4D and the Q7D groups
Arm/Group | N8-GP Prophylaxis | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Participants
  After approximately 25 months: number analyzed (Participants) | 58 | 7
  After approximately 25 months: Yes | 19 | 2
  After approximately 25 months: No | 39 | 5
  Month 25 to 80: number analyzed (Participants) | 18 | 1
  Month 25 to 80: Yes | 5 | 1
  Month 25 to 80: No | 13 | 0

48. Secondary Outcome: Number of Bleeds Using Pain Medication
Description: The mean number of bleeds using pain medication in the main phase of the study (approximately 19 months) were reported.
Time Frame: After approx 19 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Number of bleeds
Groups:
- N8-GP 50 U/kg Prophylaxis Q4D:: Participants who were on prophylaxis treatment with N8-GP in the main phase and had 0-2 bleeding episodes during the last 6 months before entering the extension phase, were included in this arm. Participants received one single bolus dose of 50 U/kg BW of N8-GP administered IV every 4th day (96 hours) or twice weekly (at investigator's discretion). The dose was adjusted to ensure a trough level of >1% FVIII:C activity in this arm. The dose was based on phase 1 data from the NN7088-3776 trial in order to ensure a trough level of >1% FVIII:C activity in the majority of participants in the prophylaxis arm.
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D: | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Number of bleeds | 0.1 (0.4) | 0.5 (1.4)

49. Secondary Outcome: Number of Adverse Events Reported During the Trial Period: After Approximately 19 Months
Description: All presented adverse events (AEs) are treatment-emergent. A treatment-emergent adverse event was defined as an event with onset after first N8-GP administration.
Time Frame: After approx 19 months
Population: Results are based on the SAS. SAS comprised all participants exposed to N8-GP in this trial.
Measure: Number; unit: Number of adverse events
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 175 | 12
Number of adverse events | 423 | 51

50. Secondary Outcome: Number of Adverse Events Reported During the Trial Period: After Approximately 25 Months
Description: as for outcome 49
Time Frame: After approx. 25 months
Population: Results are based on the SAS. SAS comprised all participants exposed to N8-GP in this trial.
Measure: Number; unit: Number of adverse events
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 175 | 38 | 12
Number of adverse events | 701 | 71 | 75

51. Secondary Outcome: Number of Adverse Events Reported During the Trial Period: After Approximately 80 Months
Description: The number of adverse events observed during the study after approximately 80 months was reported.
Time Frame: After approximately 80 months
Population: Results are based on the SAS. SAS comprised all participants exposed to N8-GP in this trial.
Measure: Number; unit: Number of adverse events
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
Number of adverse events | 1326 | 369 | 132

52. Secondary Outcome: Number of Serious Adverse Events Reported During the Trial Period: After Approximately 19 Months
Description: All presented serious adverse events (SAEs) are treatment-emergent. A treatment-emergent adverse event was defined as an event with onset after first N8-GP administration.
Time Frame: After approximately 19 months
Population: Results are based on the SAS. SAS comprised all participants exposed to N8-GP in this trial.
Measure: Number; unit: Number of serious adverse events
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 175 | 12
Number of serious adverse events | 13 | 4

53. Secondary Outcome: Number of Serious Adverse Events Reported During the Trial Period: After Approximately 25 Months
Description: as for outcome 52
Time Frame: After approximately 25 months
Population: Results are based on the SAS. SAS comprised all participants exposed to N8-GP in this trial.
Measure: Number; unit: Number of serious adverse events
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 175 | 61 | 12
Number of serious adverse events | 27 | 1 | 4

54. Secondary Outcome: Number of Serious Adverse Events Reported During the Trial Period: After Approximately 80 Months
Description: as for outcome 52
Time Frame: After approximately 80 months
Population: Results are based on the SAS. SAS comprised all participants exposed to N8-GP in this trial.
Measure: Number; unit: Number of serious adverse events
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 75 U/kg Prophylaxis Q7D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 61 | 12
Number of serious adverse events | 39 | 16 | 8

55. Secondary Outcome: Change in Blood Pressure: After Approximately 19 Months
Description: The mean change in the systolic and diastolic blood pressure values of participants was reported. The summary of change was based on individual changes observed at visit 13 (approximately 19 months) from visit 2a pre-dose (Month 0).
Time Frame: After approximately 19 months
Population: Results were based on the SAS. SAS comprised all participants exposed to N8-GP in this trial. Number analysed = Number of participants with available data for respective arm.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
mmHg
  Systolic blood pressure: number analyzed (Participants) | 19 | 3
  Systolic blood pressure | 6.8 (9.5) | 1.3 (20.5)
  Diastolic blood pressure: number analyzed (Participants) | 19 | 3
  Diastolic blood pressure | 3.3 (8.9) | 9.0 (5.2)

56. Secondary Outcome: Change in Blood Pressure: After Approximately 25 Months
Description: The mean change in the systolic and diastolic blood pressure values of participants was reported. The summary of change was based on individual changes observed at visit 17 (approximately month 25) from visit 13 (approximately month 19).
Time Frame: After approximately 19 and 25 months
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
mmHg
  Systolic blood pressure: number analyzed (Participants) | 104 | 7
  Systolic blood pressure | -1.337 (13.1) | -6.000 (9.5)
  Diastolic blood pressure: number analyzed (Participants) | 104 | 7
  Diastolic blood pressure | 0.337 (10.8) | 2.000 (5.9)

57. Secondary Outcome: Change in Blood Pressure: After Approximately 80 Months
Description: Change in the blood pressure was not calculated in the extension phase 2 of the study since participants were allowed to change from Q4D to Q7D and vice versa.
Time Frame: After approximately 80 months
Population: Data were not collected for this outcome measure.
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 0 | 0

58. Secondary Outcome: Change in Pulse: After Approximately 19 Months
Description: The mean change in the pulse values of participants was reported. The summary of change was based on individual changes observed at visit 13 (approximately 19 months) from visit 2a pre-dose (Month 0).
Time Frame: After approximately 19 months
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Beats per min
Groups:
- N8-GP 50 U/kg Prophylaxis Q4D: Participants in this arm received one single bolus dose of 50 U/kg BW of N8-GP administered intravenously (IV) every 4th day (96 hours) or twice weekly (investigator's discretion). The dose was adjusted to ensure a trough level of >1% FVIII:C activity in this arm.
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Beats per min | 5.3 (11.2) | 10.3 (4.6)

59. Secondary Outcome: Change in Pulse: After Approximately 25 Months
Description: The mean change in the pulse values of participants was reported. The summary of change was based on individual changes observed at visit 17 (approximately month 25) from visit 13 (approximately month 19).
Time Frame: After approximately 25 months
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Beats per min
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Beats per min | -0.644 (10.7) | 3.143 (8.2)

60. Secondary Outcome: Change in Pulse: After Approximately 80 Months
Description: Change in pulse was not calculated in the extension phase 2 of the study since participants were allowed to change from Q4D to Q7D and vice versa.
Time Frame: After approximately 80 months
Population: Data were not collected for this outcome measure.
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 0 | 0

61. Secondary Outcome: Change in Body Temperature: After Approximately 19 Months
Description: The mean change in the body temperature values of participants was reported. The summary of change was based on individual changes observed at visit 13 (approximately 19 months) from visit 2a pre-dose (Month 0).
Time Frame: After approximately 19 months
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Degree celcius
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Degree celcius | 0.0 (0.4) | -0.1 (0.2)

62. Secondary Outcome: Change in Body Temperature: After Approximately 25 Months
Description: The mean change in the body temperature (C) values of participants was reported. The summary of change was based on individual changes observed at visit 17 (approximately month 25) from visit 13 (approximately month 19).
Time Frame: After approximately 25 months
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Degree celcius
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Degree celcius | -0.079 (0.3) | -0.086 (0.6)

63. Secondary Outcome: Change in Body Temperature: After Approximately 80 Months
Description: Change in body temperature was not calculated in the extension phase 2 of the study since participants were allowed to change from Q4D to Q7D and vice versa.
Time Frame: After approximately 80 months
Population: Data were not collected for this outcome measure.
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 0 | 0

64. Secondary Outcome: Change in Respiratory Rate: After Approximately 19 Months
Description: The mean change in the respiratory rate values of participants was reported. The summary of change was based on individual changes observed at visit 13 (approximately 19 months) from visit 2a pre-dose (Month 0).
Time Frame: After approximately 19 months
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Breaths/min
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Breaths/min | -0.2 (1.9) | -2.3 (2.1)

65. Secondary Outcome: Change in Respiratory Rate: After Approximately 25 Months
Description: The mean change in the respiratory rate (breaths/min) values of participants was reported. The summary of change was based on individual changes observed at visit 17 (approximately month 25) from visit 13 (approximately month 19).
Time Frame: After approximately 25 months
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Breaths/min
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 177 | 12
Breaths/min | -0.067 (2.1) | -0.857 (2.5)

66. Secondary Outcome: Change in Respiratory Rate: After Approximately 80 Months
Description: Change in respiratory rate was not calculated in the extension phase 2 of the study since participants were allowed to change from Q4D to Q7D and vice versa.
Time Frame: After approximately 80 months
Population: Data were not collected for this outcome measure.
Arm/Group | N8-GP 50 U/kg Prophylaxis Q4D | N8-GP 20-75 U/kg On-demand
Number analyzed (Participants) | 0 | 0

67. Secondary Outcome: FVIII Activity 30 Min Post -Injection (C30min)
Description: FVIII plasma activity was measured after 30 mins of injection. This was measured at two time points Visit 2a (Week 0) and visit 7 (Week 28) during the Main Phase of the study. Chromogenic assay was performed with normal human plasma (NHP) as a calibrator
Time Frame: Week 0, week 28
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Groups:
- Pharmacokinetics Assessment Arm: Patients participating in the pharmacokinetic assessments received a single i.v. bolus injection of 50 U/kg BW of N8-GP at Visit 2a (Week 0) and at Visit 7 (Week 28). The PK sessions were 4 days long and with multiple site visits. After completion of the PK sessions the patients continued treatment in the prophylaxis arm with the next visit in line. Patients must not have received current FVIII product for at least 4 days prior to the PK session at Visit 2a (Week 0) and N8-GP for at least 7 days prior to the PK session at Visit 7 (Week 28).
Arm/Group | Pharmacokinetics Assessment Arm
Number analyzed (Participants) | 24
IU/mL
  Week 0: number analyzed (Participants) | 20
  Week 0 | 1.524 (22.65)
  Week 28: number analyzed (Participants) | 20
  Week 28 | 1.601 (16.24)

68. Secondary Outcome: Incremental Recovery (Single Dose and Steady State)
Description: Incremental recovery was defined as the dose-normalised activity recorded 30 min after end of injection. This was measured at two time points Visit 2a (Week 0) and visit 7 (Week 28) during the Main Phase of the study. Chromogenic assay was performed with normal human plasma (NHP) as a calibrator.
Time Frame: Week 0, week 28
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [(U/mL)/(IU/kg)]
Arm/Group | Pharmacokinetics Assessment Arm
Number analyzed (Participants) | 24
[(U/mL)/(IU/kg)]
  Week 0: number analyzed (Participants) | 20
  Week 0 | 0.031 (22.16)
  Week 28: number analyzed (Participants) | 20
  Week 28 | 0.034 (17.60)

69. Secondary Outcome: Trough Level (Single Dose and Steady State)
Description: Trough level was defined as the plasma FVIII activity recorded immediately before next dose is given. This was measured at two time points Visit 2a (Week 0) and visit 7 (Week 28) during the Main Phase of the study. Chromogenic assay was performed with normal human plasma (NHP) as a calibrator.
Time Frame: Week 0, week 28
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Pharmacokinetics Assessment Arm
Number analyzed (Participants) | 24
IU/mL
  Week 0: number analyzed (Participants) | 20
  Week 0 | 0.032 (138.3)
  Week 28: number analyzed (Participants) | 20
  Week 28 | 0.035 (138.4)

70. Secondary Outcome: Area Under the Curve (AUC0-inf)
Description: Area under the plasma activity versus time profile from time zero to infinity (AUC0-inf) was measured at two time points Visit 2a (Week 0) and visit 7 (Week 28) during the Main Phase of the study. It is the measure of total plasma exposure. Chromogenic assay was performed with normal human plasma (NHP) as a calibrator.
Time Frame: Pre dose and 30 min, 1, 4, 12, 24, 48, 72 and 96 hours post dose at week 0 and week 28
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*h/mL
Arm/Group | Pharmacokinetics Assessment Arm
Number analyzed (Participants) | 24
IU*h/mL
  Week 0: number analyzed (Participants) | 20
  Week 0 | 39.77 (34.41)
  Week 28: number analyzed (Participants) | 20
  Week 28 | 41.44 (30.09)

71. Secondary Outcome: Area Under the Curve (AUC0-t)
Description: Area under the plasma activity versus time profile from time zero to the last measurable activity (AUC0-t) was measured at two time points Visit 2a (Week 0) and visit 7 (Week 28) during the Main Phase of the study. Chromogenic assay was performed with normal human plasma (NHP) as a calibrator.
Time Frame: Pre dose and 30 min, 1, 4, 12, 24, 48, 72 and 96 hours post dose at week 0 and week 28
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*h/mL
Arm/Group | Pharmacokinetics Assessment Arm
Number analyzed (Participants) | 24
IU*h/mL
  Week 0: number analyzed (Participants) | 20
  Week 0 | 38.31 (33.22)
  Week 28: number analyzed (Participants) | 20
  Week 28 | 39.87 (28.22)

72. Secondary Outcome: Terminal Half Life (t1/2)
Description: t½ = ln(2) / λz, where λz is the terminal elimination rate constant. The terminal elimination rate constant was estimated using linear regression on the terminal part of the log(activity) versus time profile. This was measured at Visit 2a (Week 0) and visit 7 (Week 28) during the Main Phase of the study. Chromogenic assay was performed with normal human plasma (NHP) as a calibrator.
Time Frame: Pre dose and 30 min, 1, 4, 12, 24, 48, 72 and 96 hours post dose at week 0 and week 28
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | Pharmacokinetics Assessment Arm
Number analyzed (Participants) | 24
Hour (h)
  Week 0: number analyzed (Participants) | 20
  Week 0 | 18.27 (27.40)
  Week 28: number analyzed (Participants) | 20
  Week 28 | 18.18 (31.43)

73. Secondary Outcome: Clearance (CL)
Description: Total plasma clearance (CL) of drug after intravenous administration was reported. Clearance was calculated using the formula CL= Dose / AUC(0-inf). This was measured at two time points Visit 2a (Week 0) and visit 7 (Week 28) during the Main Phase of the study. Chromogenic assay was performed with normal human plasma (NHP) as a calibrator.
Time Frame: Pre dose and 30 min, 1, 4, 12, 24, 48, 72 and 96 hours post dose at week 0 and week 28
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | Pharmacokinetics Assessment Arm
Number analyzed (Participants) | 24
mL/h/kg
  Week 0: number analyzed (Participants) | 20
  Week 0 | 1.210 (33.22)
  Week 28: number analyzed (Participants) | 20
  Week 28 | 1.139 (29.24)

74. Secondary Outcome: Mean Residence Time (MRT)
Description: MRT = AUMC/AUC(0-inf), where AUMC is the area under the first moment curve, i.e. the area under the curve t∙C(t), calculated with the same method as AUC(0-inf) (linear trapezoidal method + extrapolated area). This was measured at two time points Visit 2a (Week 0) and visit 7 (Week 28) during the Main Phase of the study. Chromogenic assay was performed with normal human plasma (NHP) as a calibrator.
Time Frame: Pre dose and 30 min, 1, 4, 12, 24, 48, 72 and 96 hours post dose at week 0 and week 28
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | Pharmacokinetics Assessment Arm
Number analyzed (Participants) | 24
Hour (h)
  Week 0: number analyzed (Participants) | 20
  Week 0 | 25.12 (27.43)
  Week 28: number analyzed (Participants) | 20
  Week 28 | 24.91 (32.25)

75. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Apparent volume of distribution at steady state is a product of the mean residence time and clearance and was calculated using the formula - Vss = CL x MRT. This was measured at two time points Visit 2a (Week 0) and visit 7 (Week 28) during the Main Phase of the study. Chromogenic assay was performed with normal human plasma (NHP) as a calibrator.
Time Frame: Pre dose and 30 min, 1, 4, 12, 24, 48, 72 and 96 hours post dose at week 0 and week 28
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Pharmacokinetics Assessment Arm
Number analyzed (Participants) | 24
mL/kg
  Week 0: number analyzed (Participants) | 20
  Week 0 | 30.40 (24.18)
  Week 28: number analyzed (Participants) | 20
  Week 28 | 28.38 (19.43)

ADVERSE EVENTS:
Time Frame: From first exposure to N8-GP (week 0) to follow up visit after end of treatment in extension phase part 2. (Main phase:19 months; Extension phase 1 approximately 6 months and Extension phase 2 :approximately upto 80 months from study start).
Description: The results are based on the safety analysis set. All the presented AEs were treatment-emergent. A treatment-emergent AE was defined as an event with onset after first N8-GP administration.
Groups:
- N8-GP 50 U/kg Q4D Prophylaxis: Participants who were on prophylaxis treatment with N8-GP in the main phase and had 0-2 bleeding episodes during the last 6 months before entering the extension phase, were included in this arm. Participants received one single bolus dose of 50 U/kg BW of N8-GP administered IV every 4th day (96 hours) or twice weekly (at investigator's discretion). The dose was adjusted to ensure a trough level of >1% FVIII:C activity in this arm. The dose was based on phase 1 data from the NN7088-3776 trial in order to ensure a trough level of >1% FVIII:C activity in the majority of participants in the prophylaxis arm.
- N8-GP 75 U/kg Q7D Prophylaxis: Participants who were on prophylaxis treatment with N8-GP in the main phase and had 3+ bleeding episodes during the last 6 months before entering the extension phase, were randomised to receive one single bolus dose of 75 U/kg BW of N8-GP. Participants received one single bolus dose of 75 U/kg BW of N8-GP administered IV every 7th day (Q7D). Based on the bleeding pattern, the investigator could change the dosing frequency from Q7D to Q4D, but not vice versa. The dose was based on phase 1 data from the NN7088-3776 trial in order to ensure a trough level of >1% FVIII:C activity in the majority of participants in the prophylaxis arm.
Arm/Group | N8-GP 50 U/kg Q4D Prophylaxis | N8-GP 75 U/kg Q7D Prophylaxis | N8-GP 20-75 U/kg On-demand
All-Cause Mortality (participants affected / at risk) | 1/177 | 0/61 | 0/12
Serious Adverse Events (participants affected / at risk) | 24/177 | 7/61 | 3/12
Other Adverse Events (participants affected / at risk) | 144/177 | 50/61 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N8-GP 50 U/kg Q4D Prophylaxis (N=177) | N8-GP 75 U/kg Q7D Prophylaxis (N=61) | N8-GP 20-75 U/kg On-demand (N=12)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Factor VIII inhibition (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastric varices (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Infective spondylitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mesenteric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Skin graft infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N8-GP 50 U/kg Q4D Prophylaxis (N=177) | N8-GP 75 U/kg Q7D Prophylaxis (N=61) | N8-GP 20-75 U/kg On-demand (N=12)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 9 (12) | 3 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 12 (17) | 3 (3) | 3 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (43) | 15 (21) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 10 (11) | 3 (5) | 3 (5)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (11) | 6 (6) | 3 (3)
Blister (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 9 (9) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 5 (7) | 4 (4) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 2 (2) | 1 (1)
Citrobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 5 (5) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 11 (15) | 3 (3) | 2 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 4 (5) | 1 (2)
Dental caries (Gastrointestinal disorders) | 6 (11) | 2 (2) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 9 (9) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 17 (22) | 5 (6) | 2 (2)
Dizziness (Nervous system disorders) | 6 (7) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 5 (8) | 2 (2) | 1 (2)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 10 (10) | 2 (2) | 0 (0)
Fatigue (General disorders) | 4 (4) | 1 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Folliculitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 6 (10) | 1 (1) | 3 (5)
Gastroenteritis (Infections and infestations) | 6 (9) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 35 (79) | 13 (25) | 3 (4)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 17 (18) | 4 (5) | 0 (0)
Influenza (Infections and infestations) | 16 (22) | 6 (7) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Joint injury (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 6 (7) | 5 (6) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (14) | 4 (4) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 48 (78) | 12 (16) | 5 (12)
Nausea (Gastrointestinal disorders) | 14 (20) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 4 (5) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (14) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 9 (10) | 5 (7) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 9 (10) | 2 (2) | 0 (0)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 11 (14) | 2 (3) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 10 (12) | 5 (5) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sputum abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 3 (5) | 5 (5) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Tinea infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 10 (11) | 4 (5) | 1 (2)
Toothache (Gastrointestinal disorders) | 10 (11) | 3 (5) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 37 (59) | 9 (14) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (11) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT01480180/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT01480180/SAP_001.pdf